CLINICAL TRIAL: NCT06417892
Title: A Randomized Controlled Study of 2nd-line Treatment of Advanced G/GEJ Adenocarcinoma With Fruquintinib and Albumin-paclitaxel in Combination With or Without PD-1 Antibody in Patients Who Have Failed Treatment With PD-1 Antibody
Brief Title: Fruquintinib and Albumin-paclitaxel Combined With or Without PD-1 Antibody in 2nd-line Treatment of G/GEJ Adenocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LIN YANG, Doctor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC4594
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — spartalizumab; HMPL-013; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fruquintinib + albumin paclitaxel: Fruquintinib combined with albumin paclitaxel
  Interventions: Drug: Fruquintinib; Drug: albumin paclitaxel
- Fruquintinib + albumin paclitaxel + PD-1 antibody: Fruquintinib, albumin paclitaxel combined with PD-1 antibody
  Interventions: Drug: PD-1inhibitor; Drug: Fruquintinib; Drug: albumin paclitaxel

INTERVENTIONS:
Drug: PD-1inhibitor — PD-1 antibody was selected according to first-line drug use
  Other Names: PD-1 antibody
  Groups: Fruquintinib + albumin paclitaxel + PD-1 antibody
Drug: Fruquintinib — a small molecular anti-tumor angiogensis drug
Drug: albumin paclitaxel — a kind of cytotoxic chemotherapy drug
  Other Names: nab-paclitaxel

SUMMARY:
To explore the efficacy and safety of fruquintinib and albumin-paclitaxel combined with or without PD-1 antibody in the second-line treatment of advanced gastric/gastroesophageal junction adenocarcinoma that failed to be treated by anti-PD-1 /PD-L1 regimen

DETAILED DESCRIPTION:
This is a single-center, prospective, open, randomized controlled study of patients with advanced second-line gastric/gastroesophageal junction adenocarcinoma. The study population was pathologically confirmed advanced gastric/gastroesophageal junction adenocarcinoma, which had undergone one systemic treatment; First-line exposure to immune drugs (including PD-1 drug exposure at the stage of neoadjuvant, adjuvant, and systemic therapy); For patients with metastasis and recurrence within 6 months after the end of adjuvant/neoadjuvant system treatment, the above-mentioned treatment is first-line treatment). After patients meeting the inclusion criteria signed informed consent, the study was observed from the start of treatment until death, withdrawal of informed consent, loss of follow-up, or the end of the study.

Eligible subjects will be randomly assigned to either fruquintinib combined with albumin-paclitaxel or fruquintinib combined with albumin-paclitaxel combined with PD-1 monoclonal antibody in a 1:1 ratio. A total of 60 subjects are planned to enter the study treatment, 30 in each treatment group, and enter one of the following open treatment groups:

Group A: Fruquintinib combined with albumin-paclitaxel regimen Group B: Fruquintinib, albumin-paclitaxel combined with PD-1 antibody regimen For enrolled patients, the treating physician conducted the first visit before treatment, and the follow-up visit and the last visit after treatment began. Visits were conducted in accordance with clinical norms and there was no fixed schedule for visits. Physicians collect demographic and disease-related baseline data from medical records or at the first visit prior to treatment. Treatment-related data, including adverse events and tumor status, were collected during follow-up visits. Survival follow-up was conducted every 3 months after the end of the study, either by phone, wechat or through other doctors. The last visit recorded patient death, withdrawal of informed consent, loss of visit, or end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the informed consent;
2. Age ≥18 years old;
3. Pathologically confirmed advanced gastric/gastroesophageal junction adenocarcinoma with at least one systemic treatment;
4. Frontline experienced exposure to immune drugs (including exposure to PD-1 drugs in the neoadjuvant, adjuvant, and systemic treatment stages; For patients with metastasis and recurrence within 6 months after the end of adjuvant/neoadjuvant system treatment, the above-mentioned treatment is first-line treatment);
5. ECOG's physical condition was 0-1, and did not deteriorate within 7 days;
6. BMI≥18;
7. Expected survival ≥3 months;
8. The functions of vital organs meet the following requirements (the use of any blood components and cell growth factors is not allowed within the first 14 days of enrollment) a) Absolute neutrophil count ≥1.5×109/L, white blood cell ≥4.0×109/L; b) Platelet ≥100×109/L; c) Hemoglobin ≥90g/L; d) Total bilirubin TBIL≤1.5 times ULN; e)ALT and AST≤2.5 times ULN (up to 5 times in patients with liver metastasis); f) Urea/urea nitrogen (BUN) and creatinine (Cr) ≤1.5×ULN (and creatinine clearance (CCr) ≥ 50mL/min); g) Left ventricular ejection fraction (LVEF) ≥50%; h)Fridericia's corrected QT interval (QTcF) <470 ms. i) INR≤1.5 x ULN, APTT≤1.5 x ULN.
9. Women of childbearing age need to take effective contraceptive measures;
10. Good compliance, cooperate with follow-up;

Exclusion Criteria:

1. Failure to comply with the study protocol or study procedure;
2. Previous treatment with VEGFR inhibitors;
3. Previously received paclitaxel therapy (except for those who received paclitaxel therapy in neoadjuvant or adjuvant therapy, and the treatment ended more than 6 months after the progression of the disease);
4. Known HER-2 positive patients;
5. Receive live vaccine within 4 weeks prior to enrollment or possibly during the study period;
6. Had other malignancies within 5 years prior to enrollment, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
7. Had active autoimmune disease or history of autoimmune disease within 4 weeks prior to enrollment;
8. Previously received allogeneic bone marrow transplantation or organ transplantation;
9. Subjects who are allergic to the investigational drug or any of its adjuncts;
10. Electrolyte abnormalities identified by the investigator as clinically significant;
11. Hypertension that could not be controlled by drugs before enrollment was defined as: systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥90 mmHg;
12. Had any disease or condition affecting drug absorption before enrollment, or the patient could not take the drug orally;
13. Gastrointestinal diseases such as active ulcer of stomach and duodenum, ulcerative colitis, or active bleeding of unresectable tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by researchers before enrollment;
14. Patients with significant evidence or history of bleeding tendency (hemorrhage >30 mL within 3 months, accompanied by hematemesis, stool, and blood in the stool), hemoptysis (>5 mL of fresh blood within 4 weeks), or thromboembolic events (including stroke events and/or transient ischemic attacks) within 12 months prior to enlistment;
15. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment; Congestive heart failure New York Heart Association (NYHA) Grade >2; Ventricular arrhythmias requiring medical treatment; LVEF (left ventricular ejection fraction) <50%;
16. Active or uncontrolled severe infection (≥CTCAE v5.0 grade 2 infection);
17. Known human immunodeficiency virus (HIV) infection. A known history of clinically significant liver disease, including viral hepatitis [active HBV infection, i.e., positive HBV DNA (>1×104 copies /mL or >2000 IU/ml) must be excluded for a known hepatitis B virus (HBV) carrier; Known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL);
18. Unmitigated toxicity higher than CTCAE v5.0 grade 1 due to any previous anticancer therapy, excluding alopecia, lymphocytopenia, and oxaliplatin grade ≤2 neurotoxicity;
19. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
20. Received blood transfusion therapy, blood products and hematopoietic factors, such as albumin and granulocyte colony-stimulating factor (G-CSF), within 28 days before enrollment;
21. Any other medical condition, clinically significant metabolic abnormality, physical abnormality or laboratory abnormality, which, in the investigator's judgment, reasonably suspects that the patient has a medical condition or condition that is not suitable for the use of the investigational drug (such as having seizures and requiring treatment), or which would affect the interpretation of the study results or place the patient at high risk;
22. Urine routine indicated urinary protein ≥2+, and 24-hour urinary protein volume >1.0g;
23. The patients considered by the investigators to be unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced gastric/gastroesophageal junction adenocarcinoma who failed treatment with anti-PD-1 /PD-L1 regimen.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  Progression free survival

SECONDARY OUTCOMES:
ORR | 2 years
  Objective Remission Rate
DCR | 2 years
  Disease Control Rate
DoR | 2 years
  Duration of Remission
OS | 2 years
  overall survival
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 years
  Incidence of Treatment-Emergent Adverse Events and its degree

CONTACTS AND LOCATIONS:
Overall Officials: LIN YANG, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China